CLINICAL TRIAL: NCT05824572
Title: The Effect of Clinic Visit Audio Recordings for Self-management in Older Adults
Acronym: REPLAY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Vanderbilt University Medical Center (Other); The University of Texas Medical Branch, Galveston (Other); National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Paul J. Barr, Associate Professor, Trustees of Dartmouth College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02001844; 1R01AG074959-01A1 (NIH)
Record Dates: First submitted 2023-04-07; First posted 2023-04-21 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Diabetes
Keywords: Audio recording; Diabetes Mellitus; Patient-centered communication; Self-management; Older adults; Doctor patient communication; Technology; Multimorbidity
MeSH Terms: conditions — Diabetes Mellitus | interventions — Self-Management; Aging

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to AUDIO or UC alone using a block randomization technique with the clinician acting as the blocking variable; this strategy will ensure an equal number of patients per clinician will be randomly assigned to each study arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Audio (Active Comparator): Researchers will audio record both in-person and telehealth visits of participants in the intervention group.
  Interventions: Other: Clinic visit audio recordings for self-management in older adults
- Usual care (Placebo Comparator): Participants will receive Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Clinic visit audio recordings for self-management in older adults — The intervention is audio-recordings of primary care clinic visits that are shared with participating patients. All scheduled visits with study clinicians will be recorded and shared with patients randomized to the intervention group (AUDIO) for 12 months.
  Arms: Audio
Other: Usual Care — The Usual Care arm participants will receive After Visit Summaries (AVS) per the standard delivery at each institution
  Arms: Usual care

SUMMARY:
The objective of this study is to conduct a multisite trial evaluating the impact of adding an audio recording of clinic visits (AUDIO) to usual care in older adults with multimorbidity, including diabetes, compared to After Visit Summary (AVS) alone (Usual Care; UC).

DETAILED DESCRIPTION:
The objective of this study is to conduct a multisite trial evaluating the impact of adding an audio recording of clinic visits (AUDIO) to usual care in older adults with multimorbidity, including diabetes, compared to AVS alone (Usual Care; UC). The specific aims are: Aim 1 Conduct a three-site trial in primary care where older patients with multimorbidity including diabetes (n=336) will be randomized to receive an audio recording as well as AVS (AUDIO) versus AVS alone (UC) for all scheduled clinic visits over 12 months; patients will be assessed at baseline, 1 week, 6 months and 12 months. Applicants hypothesize (Main Effect) that: compared to those receiving UC, patients randomized to also receive audio recordings (AUDIO) of clinic visits will report a greater self-management ability (Primary Outcome), with improved quality of life, medication adherence, and satisfaction (Secondary Outcomes) at 12 months.

ELIGIBILITY:
Patients participants:

Inclusion Criteria:

* Patients who are ≥ 65 years;
* Patients with multimorbidity (i.e. patient has diabetes and one or more chronic conditions including: arthritis, asthma, atrial fibrillation, cancer, chronic obstructive pulmonary disease, heart disease, depression, heart failure, hypertension, osteoporosis, kidney disease and stroke);
* Have had two or more clinic visits in the previous 12 months;
* Plan on receiving ongoing care at the clinic for the subsequent 12 months;
* Do not have any vision or hearing problems that cannot be corrected;
* Have not recorded a clinic visit for personal use i the past 6 months.

Exclusion Criteria:

* Without capacity to consent to the project;
* With schizophrenia and other psychotic disorders, substance-use disorders, uncorrectable hearing or visual impairment or a six item screener (SIS) cognitive function score ≤ 4;
* Living in skilled nursing homes or hospice;
* Patients who have audio- recorded a clinic visit for their personal use in the previous six months;
* Patients who do not speak English or Spanish;
* Patients who lack internet access;
* Patients who (a) do not have access to a personal email, (b) do not have an email address shared with a family member or patient-identified caregiver, and (c) are not interested in creating an email account between the time they are first contacted by the study team to the time that the study team requires an email address to initiate the online recording software registration.

Clinician participants:

Inclusion criteria:

* Licensed clinician (MD including clinician residents at Dartmouth Health locations, DO, APRN, NP, PA)
* Are based at the study clinic;
* Who treat adult patients.

Exclusion criteria:

* Are trainees, e.g., fellows, medical students or residents, with the exception of clinician residents at Dartmouth Health;
* Commonly audio or video record clinic visits for patient's personal use.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-01-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Patient Activation Measure-Short Form | Patient activation at 12-months from enrollment
  The Patient Activation Measure-Short Form is a 13-item patient reported measure. Scores range from 0 (low activation) to 100 (high activation).

SECONDARY OUTCOMES:
Adherence to Refills and Medications-D (ARMS-D) | Adherence at 12-months from enrollment
  Eleven-item measure of medication adherence in diabetes. Two domains: i) Medication taking; and ii) medication refill.
Global PROMIS 10 | Global PROMIS 10 at 12 month from enrollment
  Global PROMIS (Patient-Reported Outcome Measurement Information System) is a 10-item patient reported measure with two domains: mental and physical health. Domain scores range from 4 to 20, with higher scores representing better health.
Patient Satisfaction Questionnaire-18 | Patient satisfaction at 12-months from enrollment
  Patient Satisfaction Questionnaire-18 (PSQ-18) is a patient reported measure of satisfaction. It assesses seven sub-scales of satisfaction with care with scores ranging from 1 - 5 for each. We will use the two-item domain assessing general satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Barr, PhD, Principal Investigator — Dartmouth College; Kerri L Cavanaugh, MD, Principal Investigator — Vanderbilit University Medical Center; Meredith C Masel, PhD, Principal Investigator — University Texas Medical Branch
Locations (3):
- United States (3):
  - Dartmouth-Hitchcook Manchester, Manchester, New Hampshire
  - Vanderbit University Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of results in peer-reviewed journals, access to the de-identified data for research purposes will be considered if a request is made by a qualified individual (i.e., a researcher from a research institute), IRB secured, and mutually agreed upon by the PIs. Any potential users of the data will sign an agreement that no attempt to reveal personal or private information may be made. The investigators will follow the Safe Harbour Methods outlined in the guidance regarding methods for de-identification of protected health information in accordance with the HIPAA Privacy Rule.
Supporting Information: Study Protocol
Time Frame: At the completion of data analysis
Access Criteria: Contact PI to request data